CLINICAL TRIAL: NCT02356159
Title: A Phase I/II Open Label, Dose Escalation Study of Palifermin (Kepivance) in Persons Undergoing Unrelated Donor Allogeneic Hematopoietic Cell Transplantation
Brief Title: Study of Palifermin (Kepivance) in Persons Undergoing Unrelated Donor Allogeneic Hematopoietic Cell Transplantation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Najla El Jurdi, Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 150067; 15-C-0067
Record Dates: First submitted 2015-02-04; First posted 2015-02-05 (Estimated); Results first posted 2025-06-05 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Myelodysplastic Syndromes; Hodgkin's Lymphoma; Non-Hodgkin's Lymphoma; Acute Leukemia; Multiple Myeloma
Keywords: Hematopoietic Stem Cell Transplant; Lymphoma; Leukemia; Unrelated Donors
MeSH Terms: conditions — Myelodysplastic Syndromes; Hodgkin Disease; Lymphoma, Non-Hodgkin; Multiple Myeloma; Lymphoma; Leukemia | interventions — Rituximab; fludarabine; Cyclophosphamide; Mesna; Furosemide; Tacrolimus; Cytarabine; Filgrastim; etoposide phosphate; Prednisone; Vincristine; Doxorubicin; Stem Cell Transplantation; Fibroblast Growth Factor 7; Acetaminophen; Diphenhydramine; Epinephrine; Sodium Chloride; Electrocardiography; Echocardiography; Absorptiometry, Photon; Positron-Emission Tomography; Magnetic Resonance Imaging; Spinal Puncture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1/Phase 1: Dose Escalation Arm - Palifermin (Experimental): Induction chemotherapy, then palifermin at escalating doses, then conditioning chemotherapy, then allogeneic stem cell transplant, then immunosuppression.
  Interventions: Biological: Rituximab; Drug: Conditioning chemotherapy; Drug: TMS; Drug: FLAG; Drug: EPOCH-F; Procedure: Hematopoietic stem cell transplant; Drug: Palifermin; Drug: Acetaminophen; Drug: Diphenhydramine; Drug: Prednisone; Drug: Epinephrine; Other: IV Saline; Diagnostic Test: ECG; Diagnostic Test: ECHO; Diagnostic Test: MUGA; Diagnostic Test: DEXA; Diagnostic Test: CT chest; Diagnostic Test: PET; Diagnostic Test: MRI; Procedure: BM aspirate; Procedure: BM biopsy; Procedure: Lumbar puncture
- 2/Phase II Arm - Palifermin at the Recommended Phase 2 Dose (Experimental): Induction chemotherapy, then palifermin at the recommended phase 2 dose determined in Phase 1, then conditioning chemotherapy, then allogeneic stem cell transplant, then immunosuppression.
  Interventions: Biological: Rituximab; Drug: Conditioning chemotherapy; Drug: TMS; Drug: FLAG; Drug: EPOCH-F; Procedure: Hematopoietic stem cell transplant; Drug: Palifermin; Drug: Acetaminophen; Drug: Diphenhydramine; Drug: Prednisone; Drug: Epinephrine; Other: IV Saline; Diagnostic Test: ECG; Diagnostic Test: ECHO; Diagnostic Test: MUGA; Diagnostic Test: DEXA; Diagnostic Test: CT chest; Diagnostic Test: PET; Diagnostic Test: MRI; Procedure: BM aspirate; Procedure: BM biopsy; Procedure: Lumbar puncture

INTERVENTIONS:
Biological: Rituximab — Rituximab: 375 mg/m^2 intravenous (IV) day 1 for patients with cluster of differentiation 20 (CD20)-positive disease.
  Other Names: Rituxan; Riabni; Ruxience; Truxima
Drug: Conditioning chemotherapy — Fludarabine:30 mg/m^2 per day intravenous (IV) infusion over 30 minutes, daily on days -6, -5, -4, and -3; Cyclophosphamide:1200 mg/m^2 per day IV infusion over 2 hours on Days 6, -5, -4, -3. Mesna: 1200 mg/m^2 per day IV infusion, daily on days 6, -5, -4, and -3 Furosemide: 20 mg IV flat dose on days -6, -5, -4, -3; Furosemide: 20 mg IV flat dose on days -6, -5, -4, -3.
  Other Names: Fludarabine; Cyclophosphamide; Mesna; Furosemide
Drug: TMS — Tacrolimus: 0.02 mg/kg, start day 3. Continue intravenous (IV) or by mouth (PO). Taper will begin at day +60 if no acute graft-versus-host disease (GVHD) then at day +100 and discontinue at day +180 as tolerated. Methotrexate: 5 mg/m^2 IV over 15 minutes on days 1, 3, 6, and 11. Sirolimus: 12 mg PO on days -3 to 60, followed by a taper if GVHD does not develop.
  Other Names: Tacrolimus
Drug: FLAG — Fludarabine: 25 mg/m^2 per day intravenous (IV) over 30 minutes, daily on days 1-5 Cytarabine: 2,000 mg/m^2 IV over 4 hours, on Days 1, 2, 3, 4, 5. Filgrastim: 5 mcg/kg per day subcutaneous (SC) beginning 24 hours PRIOR to initiation of chemotherapy.
  Other Names: Fludarabine; Cytarabine; Filgrastim
Drug: EPOCH-F — Fludarabine: 25 mg/m^2 per day intravenous (IV) infusion over 30 minutes, daily on days 1-4. Etoposide: 50 mg/m^2 per day continuous IV infusion over 24 hours on days 1-4. Doxorubicin: 10 mg/m^2/day continuous intravenous (CIV), days 1-4. Vincristine: 0.4 mg/m^2 per day continuous IV infusion over 24 hours daily on days 1-4.
  Cyclophosphamide: 750 mg/m^2 IV infusion over 30 minutes on day 5. Prednisone: 60 mg/m^2 per day by mouth (PO) daily on days 1-5. Filgrastim: 5 mcg/kg per day SC or IV.
  Other Names: Etoposide phosphate; Prednisone; Vincristine sulfate; Cyclophosphamide; Doxorubicin hydrochloride; Fludarabine
Procedure: Hematopoietic stem cell transplant — Hematopoietic stem cell transplant
  Other Names: HSCT
Drug: Palifermin — Escalating doses of palifermin given during transplant phase.
  Other Names: Kepivance
Drug: Acetaminophen — Before each infusion of rituximab as indicated.
  Other Names: Tylenol; Ofirmev; FeverAll
Drug: Diphenhydramine — Before each infusion of rituximab as indicated.
  Other Names: Benadryl; Banophen; Nytol
Drug: Prednisone — For engraftment syndrome.
  Other Names: Rayos; Deltasone; Prednisone Intensol
Drug: Epinephrine — Emergency medication as indicated.
  Other Names: Adrenaline
Other: IV Saline — Before each infusion of rituximab as indicated.
  Other Names: Intravenous saline
Diagnostic Test: ECG — As indicated.
  Other Names: Electrocardiogram
Diagnostic Test: ECHO — As indicated.
  Other Names: Echocardiogram
Diagnostic Test: MUGA — As indicated.
  Other Names: Multigated acquisition
Diagnostic Test: DEXA — As indicated.
  Other Names: Dual-energy X-ray absorptiometry
Diagnostic Test: CT chest — As indicated.
  Other Names: Computed tomography chest
Diagnostic Test: PET — As indicated.
  Other Names: Positron-emission tomography
Diagnostic Test: MRI — As indicated.
  Other Names: Magnetic resonance imaging
Procedure: BM aspirate — As indicated.
  Other Names: Bome marrow aspirate
Procedure: BM biopsy — As indicated.
  Other Names: Bone marrow biopsy
Procedure: Lumbar puncture — As indicated.
  Other Names: LP

SUMMARY:
Background:

- In allogeneic stem cell transplantation (SCT), stem cells are taken from a donor and given to a recipient. Sometimes the recipient's immune system destroys the donors' cells. Or donor immune cells attack the recipient's tissues, called graft-versus-host disease (GVHD). This is less likely when the recipient and donor have similar human leukocyte antigens (HLA). Researchers want to see if the drug palifermin improves the results of allogeneic SCT from HLA-matched unrelated donors.

Objective:

- To see if high doses of palifermin before chemotherapy are safe, prevent chronic GVHD, and improve immune function after transplant.

Eligibility:

- Adults 18 years of age or older with blood or bone marrow cancer with no HLA-matched sibling donor, but with a HLA-matched unrelated donor.

Description of Research Study:

* Participants will be screened with medical history, physical exam, and blood and urine tests. They will have scans and heart and lung exams.
* Before transplant, participants will:
* Have many tests and exams. These include blood tests throughout the study and bone marrow biopsy.
* Get a central line catheter if they do not have one.
* Have 1-3 rounds of chemotherapy.
* Have more tests to make sure they can have the transplant, including medical history, physical exam, blood tests, disease specific restaging.
* Get palifermin by intravenous (IV) and conditioning chemotherapy to prepare for hematopoietic stem cell transplantation (HSCT). They will get other drugs; some they will take at least 6 months.
* Participants will get the HSCT.
* After transplant, participants will:
* Be hospitalized at least 3-4 weeks.
* Monitored at least weekly for the first 100 days.
* Stay near District of Columbia (D.C). for approximately 100 days post-transplant.
* After 100 days post-transplant - visit National Institutes of Health (NIH) 5 times the first 2 years, then yearly until 5 years post-transplant.
* Additional tests/procedures may be performed to monitor safety, response to transplant, side effects.

DETAILED DESCRIPTION:
Background:

* Graft versus host disease (GVHD) and impaired immune reconstitution are major transplant complications and barriers to improving outcomes after allogeneic hematopoietic stem cell transplantation (alloHSCT) for hematologic malignancies. GVHD is initiated when donor T-cells become alloreactive against recipient major or minor histocompatibility antigens. This process may be exacerbated during the transplantation process by exposure of tissue antigens to donor T-lymphocytes after chemotherapy-induced injury.
* Palifermin, a recombinant keratinocyte growth factor-1 (KGF-1), imitates the actions of intrinsic KGF and binds to the Fibroblast growth factor (FGF) receptor 2b, which is expressed in the epidermis, oral mucosa, gastrointestinal (GI) mucosa and urothelium, thereby increasing the regenerative capacity of these tissues. Palifermin has been shown to reduce the duration and severity of oral mucositis after intensive chemo-radiotherapy and autologous HSCT for hematologic cancers and is Food and Drug Administration (FDA) approved. In pre-clinical studies, palifermin has been shown to have an effect on control of acute or chronic GVHD and immune reconstitution after alloHSCT. However, subsequent clinical studies in alloHSCT indicate that the dose and schedule of palifermin as currently

used in humans does not optimize its activity in terms of prevention of GVHD or thymus recovery following alloHSCT.

- We hypothesize that higher doses of palifermin in the immediate pre alloHSCT conditioning setting will lead to enhanced thymopoiesis, decreased chronic GVHD, and improved immune reconstitution. A dose escalation study is necessary to determine safe dosing levels in persons undergoing alloHSCT.

Objectives:

* The primary objective of the phase I portion is to assess the safety and tolerability of the administration of the recombinant keratinocyte growth factor (KGF) palifermin in alloHSCT using unrelated donor peripheral blood stem cells.
* The primary objective of the phase II portion is to determine the incidence of severe chronic GVHD after the addition of palifermin to TMS (tacrolimus, methotrexate and sirolimus) based GVHD prophylaxis delivered in the identical fashion to the NCI 07-C-0195 study.

Eligibility:

* Adults (greater than or equal to 18 years) with advanced or high-risk hematologic malignancies (including acute myeloid leukemia (AML), acute lymphoblastic leukemia (ALL), myelodysplastic syndrome (MDS), chronic lymphocytic leukemia (CLL), non-Hodgkin lymphoma (NHL), Hodgkin lymphoma (HL), chronic myeloid leukemia (CML), multiple myeloma, and myeloproliferative neoplasm (MPN) who lack a suitable human leukocyte antigens (HLA)-matched sibling donor.
* An unrelated donor matched at a minimum of 8 alleles (HLA-A,-B,-C, and major histocompatibility complex, class II, DR beta 1 (DRB1) by high-resolution typing, identified through the National Marrow Donor Program.
* Karnofsky greater than or equal to 60 and acceptable organ functions.

Design:

* Patients will receive disease-specific induction chemotherapy etoposide phosphate, prednisone, vincristine sulfate, cyclophosphamide, and doxorubicin hydrochloride with fludarabine and rituximab (EPOCH-F/R or fludararbine, ara-c, granulocyte colony-stimulating factor (FLAG) prior to transplant as needed for disease control and immune depletion.
* All patients will receive an identical conditioning regimen consisting of cyclophosphamide 1200 mg/m^2/day intravenous (IV) for 4 days and fludarabine 30 mg/m^2/day for 4 days (transplant days -6 to -3).
* All patients will receive a peripheral blood stem cell product from an unrelated donor matched at HLA-A, -B, -C, -DRB1 (8/8) by high-resolution typing.
* Palifermin will be administered in a phase 1, open label design with the following proposed schedule:

  * Dose level 1: 180 mcg/kg on day -7
  * Dose level 2: 360 mcg/kg on day -7
  * Dose level 3: 540 mcg/kg on day -7
  * Dose level 4: 720 mcg/kg on day -7
* The phase I portion will be conducted in a standard 3+3 design; the maximum possible number of patients accrued to this portion will be 24.
* The maximum tolerated dose (MTD) from the phase I portion of the study will be used to conduct a phase II study. Total accrual on the phase II study will be 27 patients, including 3-6 patients treated at the MTD in the phase I portion of the study

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients meeting below eligibility criteria are eligible to receive suitable disease specific therapy for the purposes of disease control while the donor search takes place

* The patient is greater than or equal to 18 years of age.
* Ability of subject to understand and the willingness to sign a written informed consent document.
* Karnofsky performance score >= 60.
* No suitable HLA matched sibling donor is available, and the patient has one or more potentially suitable HLA matched unrelated donor(s) in the National Marrow Donor Registry or other available registry.
* The evaluation of donors shall be in accordance with existing National Marrow Donor Program (NMDP) Standard Policies and Procedures
* HLA-matched donors are defined by allele matching at HLA-A, -B, -C,
* There is a high likelihood that the patient, in the opinion of the principal investigator (PI) or lead associate investigator (LAI), will meet the research phase eligibility criteria and proceed to transplant after induction phase therapy is completed.
* Diagnosis of hematologic malignancy meeting at least one of the disease status criteria outlined in the table below. Diagnoses must be confirmed by the National Cancer Institute (NCI) laboratory of pathology.
* Recipients with acute myeloid leukemia (AML) in first complete remission (CR1) must have one of the following:
* Adverse cytogenetics (as evaluated by history) as defined as complex karyotype (> 3 abnormalities); inv(3) or t(3;3); t(6;9); t(6;11); monosomy 7; trisomy 8, alone or with an abnormality other than t(8;21), t(9;11), inv(16) or t(16;16); or t(11;19)(q23;p13.1) or adverse-risk per European LeukemiaNet (ELN) 2017 criteria.
* Intermediate-risk disease, such as cytogenetically normal AML (CN-AML) with mutations in FMS-like tyrosine kinase 3 (FLT3), DNA methyl transferase 3A (DMNT3A), or additional sex coombs like 1 (ASXL1) or per ELN 2017 criteria.
* Primary induction failure, defined as failure to achieve CR with primary induction chemotherapy.
* Secondary AML, defined as AML related to antecedent myeloid neoplasm or cytotoxic chemotherapy.
* Hyperleukocytosis, white blood cell (WBC) > 100,000, at diagnosis.
* Recipients with ALL in CR1 must have one of the following:
* Adverse cytogenetics defined as translocations involving t(4;11), t(1;19), t(8;14), 11q23, t(9;22) or bcr-abl rearrangement, Philadelphia chromosomelike (Ph-like ALL), or complex cytogenetic abnormalities.
* Presence of minimal residual disease using multicolor flow cytometry or other analytic technique after primary induction chemotherapy.
* Primary induction failure, defined as failure to achieve complete remission (CR) with primary induction chemotherapy.
* Recipients with myelofibrosis must have at least 2 of the following features, or be Dynamic International Prognostic Scoring System (DIPSS) intermediate-2 or high risk:
* Hemoglobin < 10 g/dl, or > 10 g/dl with transfusion dependence.
* WBC < 4,000 or > 30,000/mm^3 or requires cytoreductive therapy to maintain WBC < 30,000/mm^3.
* Abnormal cytogenetics.
* Patients with lymphoma must ideally have at least stable disease from last therapy however if the PI or LAI believes there is a high likelihood of response to induction chemotherapy (EPOCH-F+/R), then the patient may be enrolled on the induction phase arm. For enrollment on the research phase arm, the patient must have at lease stable disease which is defined as:
* Absence of disease progression for at least 8 weeks after previous therapy or 12 weeks after autologous transplantation.
* Patients who are less than 8 weeks from previous therapy or 12 weeks from autologous transplantation may participate in the study at the discretion of the PI or LAI as long as they do not have progressive disease.
* Multiple myeloma in complete remission is defined as per Dr. Brian G.M. Durie (Durie BG) et al.
* Negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and <=5% plasma cells in the bone marrow. CR requires two consecutive assessments by serum and urine immunofixation made at any time prior to enrollment. CR also requires no known evidence of progressive or new bone lesions if radiographic studies are performed. Confirmation with repeat bone marrow is not needed.
* The recipient has acceptable end organ function as defined by:
* Diffusing capacity for carbon monoxide (DLCO) > 50% of the expected value (using United States of America (USA)-Information Technology Service (ITS)-National Institutes of Health (NIH) equation) when corrected for Hgb (DLCO Adj.)
* 24hr creatinine clearance or calculated (using the Cockcroft-Gault formula) creatinine clearance > 60 ml/min/1.73 (induction phase only)
* Left ventricular ejection fraction > 45%
* Serum total bilirubin less than 2.5 mg/dl, and serum alanine aminotransferase (ALT) and aspartate transferase (AST) values less than or equal to 2.5 times the upper limit of normal. Patients with elevations of serum total bilirubin up to 10 mg/dl and/or ALT or AST up to 10 times the upper limit of normal may be considered for participation if such elevations are thought to be due to liver involvement by malignancy. However, in these latter patients, if the bilirubin (BR) level does not decrease to less than or equal to 2.5 mg/dl, or AST/ALT do not decrease to less than or equal to 2.5 times the upper limit of normal after induction chemotherapy, eligibility for the transplant (research) phase will be at the discretion of the principal investigator (PI).
* Patients who are hepatitis B core antibody positive and or have positive hepatitis B surface antigen will require hepatology consultation. The risk/benefit profile of transplant and hepatitis B will be discussed with the patient and eligibility determined by the PI or the LAI.
* Patient may have a hepatitis C infection. However, each patient will require a hepatology consultation. The risk/benefit profile of transplant and hepatitis C will be discussed with the patient and eligibility determined by the PI or the LAI.
* Palifermin has had embryotoxic and fetotoxic effects in animal studies. For this reason and because the other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of active study therapy. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

Research Phase Inclusion Criteria:

Verification of donor eligibility (clearance must be received from the NMDP)

* Donors are evaluated by NMDP affiliated donor centers per NMDP Standards.

  * Donors who are medically suitable, but ineligible by Food and Drug Administration (FDA) guidelines may still donate peripheral blood stem cells (PBSC) with documentation of urgent medical need by the PI.
  * Patients who receive stem cell products from ineligible donors will be informed of any increase in risk of transfusion-related diseases prior to initiation of conditioning chemotherapy.
* Donors who are ineligible or unwilling to donate bone marrow will not be eligible to donate to study recipients. However, in the event that the patient has already begun conditioning chemotherapy and a donor PBSC collection is terminated early for donor-related medical concerns, a bone marrow graft may be infused. Should this occur, the recipient will continue to be managed on this protocol for all transplant-related care and complications. Patient will stay on study, but clinical outcomes will not be eligible for the statistics and end point calculations.
* Inadequate stem cell collection from the selected donor is defined as less than or equal to 2 x 10^6 cluster of differentiation 34 (CD34+) cells/kg. In most cases, donor cell collections are infused fresh. If a fresh collection is found to have an inadequate cell count, the cells will still be infused, but the recipient will be removed from the study and managed clinically for all transplant related care and complications on this protocol. If the patient fails to engraft, the donor may be requested for a second collection or an emergency bone marrow harvest at the discretion of the PI and NMDP Medical Director. In the event of an inadequate collection obtained prior to patient conditioning, the donor may be asked to donate a second time, or another eligible donor may be requested.
* Renal and hepatic function continues to meet eligibility criteria, reassessed as follows:

  * 24-hour creatinine clearance or calculated (using the Cockcroft-Gault formula) creatinine clearance > 60 mL/min/1.73 m^2 (induction phase only)
  * (((140-age)*mass(kg))/(72*serum creatinine (mg/dL))) x 1.73 m^2/patients body surface area (BSA)
  * If the patient is female, multiply the above by 0.85
  * In patients with suspected liver disease, bilirubin must be less than or equal to 2.5 mg/dL, AST and ALT must be less than or equal to 2.5 times institutional upper limit of normal (ULN)
* The malignancy must be restaged prior to research phase and must not have progressed during induction chemotherapy (stable disease or better). Persons with acute leukemia, myelodysplastic syndrome (MDS)/refractory anemia with excess blasts (RAEB)-I or II or chronic myeloid leukemia (CML) with previous accelerated or blast phase must have <5% blasts in the bone marrow. Persons with chronic phase CML may have up to 10% blasts in the bone marrow.

EXCLUSION CRITERIA (applies to all phases of this protocol):

* Active infection that is not responding to antimicrobial therapy.
* Active central nervous system (CNS) involvement by malignancy (patients with known positive cerebrospinal fluid (CSF) cytology or parenchymal lesions visible by computed tomography (CT) or magnetic resonance imaging (MRI).
* Previous other malignancies unless they have undergone curative intent therapy for that malignancy and (1) have had no evidence of that disease for 5 years, and/or (2) be deemed at low risk for recurrence (less than or equal to 20% at 5 years).
* Human immunodeficiency virus (HIV) positive patients are ineligible as allogeneic stem cell transplant is not yet a proven approach in this patient population, and patients are at increased risk of lethal infections when treated with marrow suppressive therapy.
* Pregnant women are excluded from this study because palifermin has been shown to be embryotoxic and fetotoxic in animal studies. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with palifermin, breastfeeding should be discontinued for the duration of active study therapy. These potential risks may also apply to other agents used in this study.
* History of psychiatric disorder or any other condition which may compromise compliance with transplant protocol or expose patient to unnecessary risk as determined by principal investigator or lead associate investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-09-24 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alain Mina, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - National Marrow Donor Program, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI).

REFERENCES:
- [Derived] Schulz E, Curtis LM, Holtzman NG, Steinberg SM, Wloka K, Ostojic A, Mina A, El Jurdi N, Pirsl F, Carpenter A, Golagha M, Sirajuddin A, Heller T, Shaffer BC, Hakim FT, Rubin JS, Gress RE, Pavletic SZ. Phase 1/2 study of high-dose palifermin for GVHD prophylaxis in patients undergoing HLA-matched unrelated donor HCT. Blood. 2025 Aug 21;146(8):944-950. doi: 10.1182/blood.2024028303. PMID 40331908
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-C-0067.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I Palifermin Dose Level 1: 180 mcg/kg Intravenous (IV) on Day-7; Phase I Palifermin Dose Level 2: 360 mcg/kg Intravenous (IV) on Day-7; Phase I Palifermin Dose Level 3: 540 mcg/kg Intravenous (IV) on Day-7; Phase I Palifermin Dose Level 4: 720 mcg/kg Intravenous (IV) on Day-7: Induction chemotherapy, then palifermin at escalating doses, then conditioning chemotherapy, then allogeneic stem cell transplant, then immunosuppression.
- Phase 2 Palifermin 720 mcg/kg Intravenous (IV) Dose: Induction chemotherapy, then palifermin at the recommended phase 2 dose (RP2D) determined in Phase 1, then conditioning chemotherapy, then allogeneic stem cell transplant, then immunosuppression.
- Participants Enrolled But Not Treated on the Research Phase (Palifermin + Transplant).: Participants were enrolled but not treated on the Research Phase (Palifermin + transplant).
Period: Total Enrolled
Arm/Group | Phase I Palifermin Dose Level 1: 180 mcg/kg Intravenous (IV) on Day-7 | Phase I Palifermin Dose Level 2: 360 mcg/kg Intravenous (IV) on Day-7 | Phase I Palifermin Dose Level 3: 540 mcg/kg Intravenous (IV) on Day-7 | Phase I Palifermin Dose Level 4: 720 mcg/kg Intravenous (IV) on Day-7 | Phase 2 Palifermin 720 mcg/kg Intravenous (IV) Dose | Participants Enrolled But Not Treated on the Research Phase (Palifermin + Transplant).
Started | 6 | 3 | 3 | 3 | 16 | 3
Eligible for Induction Phase | 5 | 2 | 3 | 2 | 2 | 2
Eligible for Research Phase | 6 | 3 | 3 | 3 | 16 | 1
Completed | 6 | 3 | 3 | 3 | 16 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Induction Phase (Ph)
Arm/Group | Phase I Palifermin Dose Level 1: 180 mcg/kg Intravenous (IV) on Day-7 | Phase I Palifermin Dose Level 2: 360 mcg/kg Intravenous (IV) on Day-7 | Phase I Palifermin Dose Level 3: 540 mcg/kg Intravenous (IV) on Day-7 | Phase I Palifermin Dose Level 4: 720 mcg/kg Intravenous (IV) on Day-7 | Phase 2 Palifermin 720 mcg/kg Intravenous (IV) Dose | Participants Enrolled But Not Treated on the Research Phase (Palifermin + Transplant).
Started | 5 | 2 | 3 | 2 | 2 | 2
Completed | 5 | 2 | 3 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Research Ph, Ph I Dose Level 180mcg/kg
Arm/Group | Phase I Palifermin Dose Level 1: 180 mcg/kg Intravenous (IV) on Day-7 | Phase I Palifermin Dose Level 2: 360 mcg/kg Intravenous (IV) on Day-7 | Phase I Palifermin Dose Level 3: 540 mcg/kg Intravenous (IV) on Day-7 | Phase I Palifermin Dose Level 4: 720 mcg/kg Intravenous (IV) on Day-7 | Phase 2 Palifermin 720 mcg/kg Intravenous (IV) Dose | Participants Enrolled But Not Treated on the Research Phase (Palifermin + Transplant).
Started | 6 | 0 | 0 | 0 | 0 | 1
Palifermin | 6 | 0 | 0 | 0 | 0 | 0
Conditioning Chemotherapy | 6 | 0 | 0 | 0 | 0 | 0
Transplant | 6 | 0 | 0 | 0 | 0 | 0
Immunosuppression Graft Versus Host Disease (GVHD) Prophylaxis | 6 | 0 | 0 | 0 | 0 | 0
Completed | 6 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Not completed — No longer eligible for research phase | 0 | 0 | 0 | 0 | 0 | 1
Period: Research Ph, Ph I Dose Level 2 360mcg/kg
Arm/Group | Phase I Palifermin Dose Level 1: 180 mcg/kg Intravenous (IV) on Day-7 | Phase I Palifermin Dose Level 2: 360 mcg/kg Intravenous (IV) on Day-7 | Phase I Palifermin Dose Level 3: 540 mcg/kg Intravenous (IV) on Day-7 | Phase I Palifermin Dose Level 4: 720 mcg/kg Intravenous (IV) on Day-7 | Phase 2 Palifermin 720 mcg/kg Intravenous (IV) Dose | Participants Enrolled But Not Treated on the Research Phase (Palifermin + Transplant).
Started | 0 | 3 | 0 | 0 | 0 | 0
Palifermin | 0 | 3 | 0 | 0 | 0 | 0
Conditioning Chemotherapy | 0 | 3 | 0 | 0 | 0 | 0
Transplant | 0 | 3 | 0 | 0 | 0 | 0
Immunosuppression Graft Versus Host Disease (GVHD) Prophylaxis | 0 | 3 | 0 | 0 | 0 | 0
Completed | 0 | 3 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Research Ph, Ph I Dose Level 3 540mcg/kg
Arm/Group | Phase I Palifermin Dose Level 1: 180 mcg/kg Intravenous (IV) on Day-7 | Phase I Palifermin Dose Level 2: 360 mcg/kg Intravenous (IV) on Day-7 | Phase I Palifermin Dose Level 3: 540 mcg/kg Intravenous (IV) on Day-7 | Phase I Palifermin Dose Level 4: 720 mcg/kg Intravenous (IV) on Day-7 | Phase 2 Palifermin 720 mcg/kg Intravenous (IV) Dose | Participants Enrolled But Not Treated on the Research Phase (Palifermin + Transplant).
Started | 0 | 0 | 3 | 0 | 0 | 0
Palifermin | 0 | 0 | 3 | 0 | 0 | 0
Conditioning Chemotherapy | 0 | 0 | 3 | 0 | 0 | 0
Transplant | 0 | 0 | 3 | 0 | 0 | 0
Immunosuppression Graft Versus Host Disease (GVHD) Prophylaxis | 0 | 0 | 3 | 0 | 0 | 0
Completed | 0 | 0 | 3 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Research Ph, Ph I Dose Level 4 720mcg/kg
Arm/Group | Phase I Palifermin Dose Level 1: 180 mcg/kg Intravenous (IV) on Day-7 | Phase I Palifermin Dose Level 2: 360 mcg/kg Intravenous (IV) on Day-7 | Phase I Palifermin Dose Level 3: 540 mcg/kg Intravenous (IV) on Day-7 | Phase I Palifermin Dose Level 4: 720 mcg/kg Intravenous (IV) on Day-7 | Phase 2 Palifermin 720 mcg/kg Intravenous (IV) Dose | Participants Enrolled But Not Treated on the Research Phase (Palifermin + Transplant).
Started | 0 | 0 | 0 | 3 | 0 | 0
Palifermin | 0 | 0 | 0 | 3 | 0 | 0
Conditioning Chemotherapy | 0 | 0 | 0 | 3 | 0 | 0
Transplant | 0 | 0 | 0 | 3 | 0 | 0
Immunosuppression Graft Versus Host Disease (GVHD) Prophylaxis | 0 | 0 | 0 | 3 | 0 | 0
Completed | 0 | 0 | 0 | 3 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase II - Maximum Tolerated Dose
Arm/Group | Phase I Palifermin Dose Level 1: 180 mcg/kg Intravenous (IV) on Day-7 | Phase I Palifermin Dose Level 2: 360 mcg/kg Intravenous (IV) on Day-7 | Phase I Palifermin Dose Level 3: 540 mcg/kg Intravenous (IV) on Day-7 | Phase I Palifermin Dose Level 4: 720 mcg/kg Intravenous (IV) on Day-7 | Phase 2 Palifermin 720 mcg/kg Intravenous (IV) Dose | Participants Enrolled But Not Treated on the Research Phase (Palifermin + Transplant).
Started | 0 | 0 | 0 | 0 | 16 | 0
Palifermin | 0 | 0 | 0 | 0 | 16 | 0
Conditioning Chemotherapy | 0 | 0 | 0 | 0 | 16 | 0
Transplant | 0 | 0 | 0 | 0 | 16 | 0
Immunosuppression Graft Versus Host Disease (GVHD) Prophylaxis | 0 | 0 | 0 | 0 | 16 | 0
Completed | 0 | 0 | 0 | 0 | 16 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are reported for participants enrolled but not treated.
Groups:
- Phase 2 Palifermin: 720 mcg/kg Intravenous (IV) Dose: Induction chemotherapy, then palifermin at the recommended phase 2 dose (RP2D) determined in Phase 1, then conditioning chemotherapy, then allogeneic stem cell transplant, then immunosuppression.
- Participants Enrolled But Not Treated on Research Phase (Palifermin + Transplant): Participants were enrolled but not treated on Research Phase (Palifermin + Transplant).
- Total: Total of all reporting groups
Arm/Group | Phase I Palifermin Dose Level 1: 180 mcg/kg Intravenous (IV) on Day-7 | Phase I Palifermin Dose Level 2: 360 mcg/kg Intravenous (IV) on Day-7 | Phase I Palifermin Dose Level 3: 540 mcg/kg Intravenous (IV) on Day-7 | Phase I Palifermin Dose Level 4: 720 mcg/kg Intravenous (IV) on Day-7 | Phase 2 Palifermin: 720 mcg/kg Intravenous (IV) Dose | Participants Enrolled But Not Treated on Research Phase (Palifermin + Transplant) | Total
Number analyzed (Participants) | 6 | 3 | 3 | 3 | 16 | 3 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 3 | 3 | 3 | 16 | 2 | 33
  >=65 years | 0 | 0 | 0 | 0 | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (10.01) | 55.67 (8.62) | 31 (10.15) | 46.33 (11.06) | 35.19 (12.5) | 61 (7) | 42.41 (14.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 0 | 0 | 6 | 1 | 11
  Male | 4 | 1 | 3 | 3 | 10 | 2 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 2 | 1 | 12 | 0 | 16
  Not Hispanic or Latino | 5 | 3 | 1 | 2 | 4 | 3 | 18
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Asian | 2 | 1 | 0 | 0 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 0 | 0 | 1
  White | 4 | 1 | 2 | 2 | 12 | 3 | 24
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 3 | 0 | 5
Region of Enrollment [Number; unit: participants]
  United States | 6 | 3 | 3 | 3 | 16 | 3 | 34

OUTCOME MEASURES:

1. Primary Outcome: Phase II: Estimated Percent of Participants Who Experienced Severe Chronic Graft Versus Host Disease (GVHD)
Description: The estimated percent of participants who experienced severe chronic graft versus host disease (GVHD) was assessed by the 1994 Consensus Conference Working Criteria. Severe GVHD is defined using the Global Staging per 2014 National Institutes of Health (NIH) Consensus Criteria for chronic GVHD.
Time Frame: 60 months
Population: The total number of participants analyzed for the primary outcome measure is 19 (16 enrolled on the phase 2 Arm and data/outcomes on the 3 participants from phase 1 treated at dose level 4).
Measure: Number (95% Confidence Interval); unit: Estimated percent of participants
Groups:
- 2/Phase II Arm - Palifermin at the Recommended Phase 2 Dose: Induction chemotherapy, then palifermin at the recommended phase 2 dose (RP2D) determined in Phase 1, then conditioning chemotherapy, then allogeneic stem cell transplant, then immunosuppression.
Arm/Group | 2/Phase II Arm - Palifermin at the Recommended Phase 2 Dose
Number analyzed (Participants) | 19
Estimated percent of participants | 6.0 [0.3 to 24.7]

2. Primary Outcome: Phase I: Maximum Tolerated Dose (MTD) of Palifermin
Description: MTD is defined as the dose level at which no more than 1 (of ≤ 6) participants who experience dose-limiting toxicity (DLT), and the dose below that at which at least 2 (of ≤ 6) participants have a DLT as a result of the drug. A DLT is non-relapse mortality before day 30 post transplantation regardless of attribution to palifermin. and non-hematologic grade 4 (life-threatening) adverse events within 14 days after treatment with palifermin possibly related to drug.
Time Frame: Approximately 30-day post-transplant
Population: All participants = (total # for phase 1).
Measure: Number; unit: mcg/kg
Groups:
- All Phase I Participants: All participants who received at least one dose of palifermin.
Arm/Group | All Phase I Participants
Number analyzed (Participants) | 15
mcg/kg | 720

3. Primary Outcome: Phase 1: Number of Participants With a Dose-limiting Toxicity (DLT)
Description: A DLT is non-relapse mortality before day 30 post transplantation regardless of attribution to palifermin. Persons who expire from malignancy related causes are not considered DLTs; and non-hematologic Common Terminology Criteria for Adverse Events (CTCAE) ≥ grade 4 adverse events (AEs), occurring within 14 days after administration of palifermin that are determined by the investigator to be at least possibly related to the study drug. An isolated laboratory value is not considered an AE unless it meets the guidelines. Note: Participants will not be removed from study therapy due to palifermin toxicity as only 1 dose is administered. DLT criteria are established only to determine dose levels for subsequent participants.
Time Frame: ≤day 30 post-transplant
Population: 15/16 participants were analyzed because 1 participant was a screen failure post induction for research phase.
Measure: Count of Participants; unit: Participants
Arm/Group | 1/Phase 1: Dose Escalation Arm - Palifermin
Number analyzed (Participants) | 15
Participants | 1

4. Other Pre Specified Outcome: Phase I and/or Phase 2: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: All adverse events, including clinically significant abnormal findings on laboratory evaluations, regardless of severity, will be followed until return to baseline or stabilization of event, up to 5 years.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Palifermin Dose Level 1: 180 mcg/kg Intravenous (IV) on Day-7 | Phase I Palifermin Dose Level 2: 360 mcg/kg Intravenous (IV) on Day-7 | Phase I Palifermin Dose Level 3: 540 mcg/kg Intravenous (IV) on Day-7 | Phase I Palifermin Dose Level 4: 720 mcg/kg Intravenous (IV) on Day-7 | Phase 2 Palifermin: 720 mcg/kg Intravenous (IV) Dose | Participants Enrolled But Not Treated on Research Phase (Palifermin + Transplant)
Number analyzed (Participants) | 6 | 3 | 3 | 3 | 16 | 3
Participants | 6 | 3 | 3 | 3 | 16 | 0

ADVERSE EVENTS:
Time Frame: All adverse events, including clinically significant abnormal findings on laboratory evaluations, regardless of severity, will be followed until return to baseline or stabilization of event, up to 5 years
Groups:
- Participants Enrolled But Not Treated on the Research Phase (Palifermin + Transplant): Participants were enrolled but not treated on Research Phase (Palifermin + Transplant).
Arm/Group | Phase I Palifermin Dose Level 1: 180 mcg/kg Intravenous (IV) on Day-7 | Phase I Palifermin Dose Level 2: 360 mcg/kg Intravenous (IV) on Day-7 | Phase I Palifermin Dose Level 3: 540 mcg/kg Intravenous (IV) on Day-7 | Phase I Palifermin Dose Level 4: 720 mcg/kg Intravenous (IV) on Day-7 | Phase 2 Palifermin: 720 mcg/kg Intravenous (IV) Dose | Participants Enrolled But Not Treated on the Research Phase (Palifermin + Transplant)
All-Cause Mortality (participants affected / at risk) | 2/6 | 2/3 | 1/3 | 1/3 | 6/16 | 0/3
Serious Adverse Events (participants affected / at risk) | 3/6 | 2/3 | 2/3 | 1/3 | 5/16 | 0/3
Other Adverse Events (participants affected / at risk) | 6/6 | 3/3 | 3/3 | 3/3 | 16/16 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Palifermin Dose Level 1: 180 mcg/kg Intravenous (IV) on Day-7 (N=6) | Phase I Palifermin Dose Level 2: 360 mcg/kg Intravenous (IV) on Day-7 (N=3) | Phase I Palifermin Dose Level 3: 540 mcg/kg Intravenous (IV) on Day-7 (N=3) | Phase I Palifermin Dose Level 4: 720 mcg/kg Intravenous (IV) on Day-7 (N=3) | Phase 2 Palifermin: 720 mcg/kg Intravenous (IV) Dose (N=16) | Participants Enrolled But Not Treated on the Research Phase (Palifermin + Transplant) (N=3)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaphylaxis (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Corneal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Corneal ulcer (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death NOS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, CMV reactivation (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, CMV infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, CMV Reactivation (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, CMV Viremia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, Specify (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — +Streptococcus Mitis (viridans Strep) 1/29/2019 blood culture
Lipase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rhinitis infective (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Palifermin Dose Level 1: 180 mcg/kg Intravenous (IV) on Day-7 (N=6) | Phase I Palifermin Dose Level 2: 360 mcg/kg Intravenous (IV) on Day-7 (N=3) | Phase I Palifermin Dose Level 3: 540 mcg/kg Intravenous (IV) on Day-7 (N=3) | Phase I Palifermin Dose Level 4: 720 mcg/kg Intravenous (IV) on Day-7 (N=3) | Phase 2 Palifermin: 720 mcg/kg Intravenous (IV) Dose (N=16) | Participants Enrolled But Not Treated on the Research Phase (Palifermin + Transplant) (N=3)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (4) | 1 (2) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Akathisia (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Allergic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bladder infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Bronchial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CPK increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Death NOS (due to disease progression) (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Per protocol death&hospitalization that are deemed to be due to disease progression & not attributable to the intervention will not be reported as a serious adverse event unless there is evidence suggesting a causal relationship (intervention/event).
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 5 (6) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Edema face (General disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 4 (4) | 0 (0)
Gastrointestinal disorders - Other, Tongue thickness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, Tongue thickness/discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 7 (16) | 0 (0)
Heart failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (7) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 4 (5) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (5) | 2 (2) | 0 (0) | 1 (1) | 7 (10) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 6 (6) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 8 (19) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, +Coronavirus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, +EBV>+2.70Log 10(intermittent) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, Acinetobacter radioresistens (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, Bacteremia; E.coli (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, Bacteremia; Mycobacterium chelonae (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, CMV (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Infections and infestations - Other, CMV + biopsy (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, CMV Reactivation (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, CMV reactivation (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Infections and infestations - Other, COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, EBV (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Infections and infestations - Other, EBV Positive (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, EBV Reactivation (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, EBV reactivation (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, Influenza B infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, Rhodotorula mucilaginosa (Yeast) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, Stenotrophomonas Maltophilia+ (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Lipase increased (Investigations) | 2 (5) | 0 (0) | 1 (1) | 2 (4) | 3 (6) | 0 (0)
Malaise (General disorders) | 1 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolism and nutrition disorders - Other, Low Vitamin D level (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (5) | 3 (4) | 1 (2) | 1 (1) | 10 (11) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nervous system disorders - Other, Presence of Chvostek sign (due to hypocalcemia) (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Oral dysesthesia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 5 (5) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 3 (3) | 3 (4) | 11 (12) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, Specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Irritation to chest when coughing (treated w/incentive spirometer Q 8 hrs.)
Rhinitis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Serum amylase increased (Investigations) | 3 (5) | 1 (1) | 1 (1) | 2 (2) | 7 (20) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Specify (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Erythema and "sunburn-like" discomfort to face, palms and soles
Skin and subcutaneous tissue disorders - Other, toxic erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Stomal ulcer (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (5) | 7 (9) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 5 (7) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-09-05): https://cdn.clinicaltrials.gov/large-docs/59/NCT02356159/Prot_SAP_002.pdf
  • Informed Consent Form (2022-05-24): https://cdn.clinicaltrials.gov/large-docs/59/NCT02356159/ICF_001.pdf